CLINICAL TRIAL: NCT02783482
Title: An Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) GC5107 in Subjects With Primary Humoral Immunodeficiency
Brief Title: Study of Immune Globulin Intravenous (Human) GC5107 in Subjects With Primary Humoral Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Parexel (Industry); Atlantic Research Group (Other)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5107B_P3
Record Dates: First submitted 2016-04-24; First posted 2016-05-26 (Estimated); Results first posted 2022-10-28 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-09

CONDITIONS: Immunologic Deficiency Syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — gamma-Globulins; Solutions; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GC5107 (Experimental): GC5107 Immune globulin intravenous (human) solution, 10% liquid
  Interventions: Biological: GC5107

INTERVENTIONS:
Biological: GC5107 — GC5107 20g/200mL, intravenously, dose of 300 - 900 mg/kg (of body weight) every 21 or 28 days for 12 months, a follow-up (3 or 4 weeks)
  Other Names: IGIV; Immune globulin intravenous (human) solution, 10% liquid

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) GC5107 in subjects with Primary Humoral Immunodeficiency (PHID).

DETAILED DESCRIPTION:
This was a prospective, open-label, single-arm, historically controlled, multicenter phase 3 study measuring the safety, efficacy and pharmacokinetics and tolerability of GC5107 in subjects with Primary Humoral Immunodeficiency disease (PHID).

Subjects received intravenous infusions of the investigational product at the same dose and interval as used for their previous Immunoglobulin intravenous (IVIG) maintenance therapy. GC5107 was administered every 21 or 28 days for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a confirmed clinical diagnosis of a Primary Humoral Immunodeficiency Disease as defined by IUIS (International Union of Immunological Societies) and require treatment with IGIV. Documented agammaglobulinemia or hypogammaglobulinemia
* Male or Female, ages 2 to 70 years
* The subject has received 300-900 mg/kg of a licensed IGIV therapy at 21 or 28 day intervals for at least 3 months prior to this study
* At least 2 documented IgG trough levels of ≥ 500 mg/dL are obtained at two infusion cycles (21 or 28 days) within 12 months prior to study enrollment

Exclusion Criteria:

* Subject has secondary immunodeficiency
* Subject was newly diagnosed with PHID and has not yet been treated with immunoglobulin
* Subject has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency or isolated IgA deficiency with known anti-IgA antibodies
* History of severe reaction or hypersensitivity to IGIV or other injectable form of IgG
* Subject has a lifetime history of at least one thrombotic event including deep vein thrombosis, cerebrovascular accident, pulmonary embolism, transient ischemic attacks, or myocardial infarction
* Subject has received blood products other than human albumin or human immunoglobulin within 12 months prior to enrollment

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (10):
  - Immuno International Research Centers, Centennial, Colorado
  - Allergy Associates of Palm Beaches PA, North Palm Beach, Florida
  - Midwest Immunology Clinic and Infusion Center, Plymouth, Minnesota
  - Optimed Infusions LLC, Columbus, Ohio
  - Oklahoma Institute of Allergy Ashma and Immunology, Oklahoma City, Oklahoma
  - Allergy Partners of North Texas Research, Dallas, Texas
  - Allergy and Asthma Specialists, Dallas, Texas
  - Pediatric Pulmonary Associates of North Texas, Frisco, Texas
  - Allergy Asthma and Immunology Clinic PA, Irving, Texas
  - Lysosomal Rare Disorder Research and Treatment Center, Inc., Fairfax, Virginia
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Queen's University - Kingston General Hospital (KGH), Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Hotel Dieu de Montreal, Montreal, Quebec
  - CHU Ste-Justine - University of Montreal, Montreal, Quebec
  - McGill University Health Centre (MUHC) - The Montreal Children's Hospital, Montreal, Quebec
  - Clinique Spécialisée en Allergie de la Capitale, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez EE, Hebert J, Ellis AK, Alpan O, Lumry WR, Shapiro R, Suez D, Mandujano JF, Wasserman RL. Efficacy, Safety and Tolerability of a New 10% Intravenous Immunoglobulin for the Treatment of Primary Immunodeficiencies. Front Immunol. 2021 Jul 8;12:707463. doi: 10.3389/fimmu.2021.707463. eCollection 2021. PMID 34305948

RESULTS

PARTICIPANT FLOW:
Groups:
- 28-day Schedule: Infusion every 28 days
- 21-day Schedule: Infusion every 21 days
Period: Overall Study
Arm/Group | 28-day Schedule | 21-day Schedule
Started | 29 | 20
Completed | 24 | 19
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- 28-day Infusion: Infusion every 28 days
- 21-day Infusion: Infusion every 21 days
- Total: Total of all reporting groups
Arm/Group | 28-day Infusion | 21-day Infusion | Total
Number analyzed (Participants) | 29 | 20 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (21.7) | 30.7 (23.2) | 37.1 (22.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 16 | 12 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 19 | 47
  Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 2 | 13
  United States | 18 | 18 | 36
Duration since first IVIG infusion [Mean (Standard Deviation); unit: years] | 8.8 (8.3) | 8.8 (6.7) | 8.8 (7.6)
IVIG dose prior to enrollment [Mean (Standard Deviation); unit: mg/kg] | 501.2 (94.0) | 592.7 (135.9) | 538.5 (120.6)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Acute Serious Bacterial Infections (SBI)
Description: The incidence of acute serious bacterial infections (aSBIs) meeting FDA guidance criteria, which includes bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscesses, and osteomyelitis/septic arthritis.
  Efficacy data is evaluated by comparing the frequency of acute serious bacterial infections per subject per year according to the FDA guideline of an upper one-sided 99% confidence limit < 1.0 per subject per year.
Time Frame: One year
Population: Intent-to-Treat (ITT) Population: Defined as of all subjects who were enrolled into the study and received any amount of the IMP. This population was used for display of demographics, disposition, and for the primary safety and efficacy analyses
Measure: Number (99% Confidence Interval); unit: Number of events per patient per year
Groups:
- 28-day Schedule: GC5107 was administered at a dose of 300-900 mg/kg (of body weight) every 28 days for 12 months of study infusions.
- 21-day Schedule: GC5107 was administered at a dose of 300-900 mg/kg (of body weight) every 21 days for 12 months of study infusions.
- Total: 28-Day schedule and 21-Day schedule
Arm/Group | 28-day Schedule | 21-day Schedule | Total
Number analyzed (Participants) | 29 | 20 | 49
Number of events per patient per year | 0.04 [NA to 0.35] — Pre-specified to only calculate the upper limit of the CI | 0 [NA to NA] — Here NA signifies that the upper limit of 99% CI was not estimable due to zero number of events | 0.02 [NA to 0.21] — Pre-specified to only calculate the upper limit of the CI

2. Primary Outcome: The Proportion of Infusions With Temporally Associated Adverse Events (TAAEs) That Occur Within 72 Hours Following an Infusion of Test Product
Description: The proportion of infusions with temporally associated adverse events occurring during or within 72 hours following infusion, whether or not they were thought to be related to GC5107
Time Frame: Within 72 hours after an infusion of GC5107
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of infusion with TAAEs
Units Other Than Participants: Total No of infusions
Arm/Group | 28-day Schedule | 21-day Schedule | Total
Number analyzed (Participants) | 29 | 20 | 49
Number analyzed (Total No of infusions) | 335 | 332 | 667
Proportion of infusion with TAAEs | 0.31 [NA to 0.40] — Pre-specified to only calculate the upper limit of the CI, meeting FDA guidance | 0.16 [NA to 0.22] — Pre-specified to only calculate the upper limit of the CI, meeting FDA guidance | 0.24 [NA to 0.31] — Pre-specified to only calculate the upper limit of the CI, meeting FDA guidance

3. Secondary Outcome: The Incidence of Infections Other Than Acute Serious Bacterial Infections
Time Frame: One year
Population: as for outcome 1
Measure: Number; unit: Numberof infections per patient per year
Arm/Group | 28-day Schedule | 21-day Schedule | Total
Number analyzed (Participants) | 29 | 20 | 49
Numberof infections per patient per year | 2.4 | 3.6 | 2.9

4. Secondary Outcome: The Number of Days Missed From Work/School/Kindergarten/Daycare, or Days Unable to Perform Normal Daily Activities Due to Infections
Description: Based on the total number of days missed from work/school/kindergarten/daycare or days unable to perform normal daily activities due to infections for each subject. Mean and SD are calculated based on weighting for the duration of data available for each subject, where duration is defined as (date of last visit - first infusion date + 1) for subjects who complete the study; and defined as (date of withdrawal - first infusion date + 1) for subjects who withdraw from the study.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 28-day Schedule | 21-day Schedule | Total
Number analyzed (Participants) | 29 | 20 | 49
Days | 2.9 (4.20) | 12.7 (26.11) | 7.1 (18.04)

5. Secondary Outcome: The Number of Days of Unscheduled Physician Visits Due to Infections
Description: Based on the total number of days of unscheduled physician visits due to infections for each subject. Mean and SD are calculated based on weighting for the duration of data available for each subject, where duration is defined as (date of last visit - first infusion date + 1) for subjects who complete the study; and defined as (date of withdrawal - first infusion date + 1) for subjects who withdraw from the study.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Groups:
- GC5107 IVIG 10%: GC5107 IVIG 10% 28-day and 21-day infusion schedule
Arm/Group | 28-day Schedule | 21-day Schedule | GC5107 IVIG 10%
Number analyzed (Participants) | 29 | 20 | 49
Days | 2.3 (4.56) | 2.4 (2.25) | 2.3 (3.75)

6. Secondary Outcome: The Number of Days of Hospitalizations Due to Infections
Description: Subject with no experience of specific event will be included in the analysis as zero incidence, zero day, or zero time duration. The mean and SD will be calculated weighting for the duration of data available for each subject.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 28-day Schedule | 21-day Schedule | Total
Number analyzed (Participants) | 29 | 20 | 49
Days | 0.1 (0.57) | 0.1 (0.46) | 0.1 (0.53)

7. Secondary Outcome: The Number of Days of Intravenous (IV) Therapeutic Antibiotics
Description: Based on the total number of days of IV therapeutic antibiotics for each subject. Mean and SD are calculated based on weighting for the duration of data available for each subject, where duration is defined as (date of last visit -first infusion date + 1) for subjects who complete the study; and defined as (date of withdrawal - first infusion date + 1) for subjects who withdraw from the study.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 28-day Schedule | 21-day Schedule | GC5107 IVIG 10%
Number analyzed (Participants) | 29 | 20 | 49
Days | 0.1 (0.57) | 0.0 (0.00) | 0.1 (0.44)

8. Secondary Outcome: The Number of Days of Oral Therapeutic Antibiotics
Description: Based on the total number of days of oral (PO) therapeutic antibiotics for each subject. Mean and SD are calculated based on weighting for the duration of data available for each subject, where duration is defined as (date of last visit - first infusion date + 1) for subjects who complete the study; and defined as (date of withdrawal - first infusion date + 1) for subjects who withdraw from the study.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 28-day Schedule | 21-day Schedule | GC5107 IVIG 10%
Number analyzed (Participants) | 29 | 20 | 49
Days | 13.3 (24.50) | 13.1 (18.38) | 13.2 (22.09)

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | GC5107 IVIG 10%
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 4/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC5107 IVIG 10% (N=49)
Influenza (Infections and infestations) | 1 (1)
Acute urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
ST elevation myocardial infarction (Cardiac disorders) | 1 (1) — Occurred after 43 weeks of GC5107 treatment and 22 days after the last infusion prior to the event, Not related to IMP
Bacterial pneumonia (Infections and infestations) | 1 (1)
Squamous cell carcinoma of base of tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GC5107 IVIG 10% (N=49)
Headache (Nervous system disorders) | 28
Nausea (Gastrointestinal disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Fatigue (General disorders) | 13
Pyrexia (General disorders) | 13
Sinusitis (Infections and infestations) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Bronchitis (Infections and infestations) | 6
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Acute sinusitis (Infections and infestations) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5
Urinary tract infection (Infections and infestations) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Viral infection (Infections and infestations) | 4
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 3
Dizziness (Nervous system disorders) | 3
Ear pain (Eye disorders) | 3
Gastroenteritis viral (Infections and infestations) | 3
Infusion site extravasation (General disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Otitis media (Infections and infestations) | 3
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Sinus headache (Nervous system disorders) | 3
Urine analysis abnormal (Investigations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT02783482/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT02783482/SAP_001.pdf